CLINICAL TRIAL: NCT05544305
Title: Digitised Home Based Care for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Associate Professor of eHealth, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PEOS-3289
Record Dates: First submitted 2022-09-01; First posted 2022-09-16 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Parkinson
Keywords: Parkinson Disease; Self-Management; Telemedicine; Artificial Intelligence
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Masking Description: No blinding will be possible in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digitised Home Based Care pathway (Experimental): The investigators have co-designed an innovative digital care pathway, Home Based Care (HBC), that delivers self-management support and clinical expertise to the patient's home, supported by digitally-enabled remote monitoring with a wrist-worn sensor, the Parkinson's Kinetograph, and digitally-delivered questionnaires, to replace the current pen-and-paper processes.
  Interventions: Other: Digital Home Based Care pathway

INTERVENTIONS:
Other: Digital Home Based Care pathway — The digital version of the pathway includes an integrated data platform with an automated patient flow management system, digitised patient-reported outcome on web-based patient portal, and AI-based automated reporting for clinical decision support.

SUMMARY:
Parkinson's disease is the world's fastest-growing neurological condition. It is a progressive neurodegenerative disorder that causes a wide range of movement-related (motor) problems (slowness, stiffness, tremor, balance difficulties) and non-motor problems (disturbances of thinking, memory, perception, mood, bladder, bowels, blood pressure). Even before the pandemic, NHS services were struggling to meet the demand for care.

To address this need for support, the investigators have co-designed an innovative digital care pathway, Home Based Care (HBC), with people with Parkinson's (PwP) and care partners (CP) to deliver self-management support and clinical expertise to the patient's home. This pathway is supported by remote monitoring with a wrist-worn sensor and questionnaires.

In this study, the investigators will be digitising this pathway so that data from a variety of sources (including the sensor, questionnaires, and patients' health records) can be combined in one place to enable more personalised care and to provide advice to support self-management of symptoms by patients.

After the investigators have set up the digitised pathway, its implementation will be evaluated with a group of 120 people with Parkinson's and their care partners and associated healthcare providers through the Plymouth Parkinson's Service. The investigators will examine participants' adoption of and engagement with the patient-facing digital platform over the course of 3 months and gather their feedback about its usability and acceptability. A smaller group of the participants will discuss their experiences in more detail to help pinpoint aspects that work well and those needing adjustment and development.

The investigators anticipate that this system will result in improved quality of life and care and increased knowledge and confidence for self-managing symptoms. The results of the study will be used to improve the digitised Home Based Care pathway. People with Parkinson's and care partners involved in the project will help guide the sharing of these results with healthcare providers and the general public.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Not resident in care home or nursing home
* Ambulant
* Have compatible smartphone/data access (access to a digital device is a necessary prerequisite of system use, and the formative usability study had success in recruiting participants with varying levels of experience with smartphones [18])
* Be fluent in English
* Normally under the care of the Parkinson's service in the participating organisation
* Participant's healthcare provider in the participating organisation consented to participate in the study
* Able and willing to provide informed consent
* Able and willing to comply with intervention requirements

Exclusion Criteria:

* Secondary cause of parkinsonism
* Significant cognitive impairment or a diagnosis of Parkinson's disease dementia
* Significant comorbidity, which in the opinion of the chief investigator would preclude safe participation in the study or protocol compliance
* Previous involvement in development or testing of the NMS Assist system
* A life expectancy of <6 months
* Living in residential care facilities
* Incapable of self-consent
* In a dependent/unequal relationship with the research or care teams or any PPI representatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Uptake | 3 months
  Rates of conversion to the digital platform
Degree of compliance with wearable sensor | 3 months
  The wearable sensors are worn on the wrist and are known as the Parkinson's Kinetograph (PKG). The PKG assess objective motor measures including bradykinesia, dyskinesia and tremor. In accordance with the HBC pathway, patients are required to wear the PKG for 6 days and nights, after which the results are analyzed by their care team. From these results, therefore, it is clear to see where the patient has complied with wearing the PKG for the allotted time frame.
Proportion of digital questionnaires completed | 3 months
  In accordance with HBC pathway, patients are required to complete a set of questionnaires covering the same time period in which they are wearing the PKG, and are responsible for assessing subjective measures. This outcome will assess compliance by examining the patients' overall compliance with the digital monitoring questionnaires by calculating how many of the questionnaires they successfully complete over the study period.
Engagement | 3 months
  Qualitative feedback about engagement from semi-structured interviews

SECONDARY OUTCOMES:
Usability scores | 3 months
  System Usability Scale, 5-point Likert scale with total scores ranging from 0-100
Patient perceptions of usability | 3 months
  Qualitative feedback about usability from semi-structured interviews
Patient perceptions of acceptability | 3 months
  Qualitative feedback about acceptability from semi-structured interviews
Cost impact | 3 months
  Preliminary evaluation of implementation costs; costs required to implement the digital HBC pathway will be compared to the costs of delivering the standard care pathway

CONTACTS AND LOCATIONS:
Overall Officials: Camille Carroll, PhD, Principal Investigator — University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the project leads and associated staff will have access to the research data and healthcare professionals participating in the study will have access only to the data from the PwP and care partners whom they are treating.